CLINICAL TRIAL: NCT00993200
Title: PerMIT: Warfarin : A Prospective Randomized Controlled Trial Comparing Usual Care Warfarin Initiation to PerMIT Pharmacogenetic Guided Warfarin Therapy
Brief Title: Personalized Medicine Interface Tool (PerMIT): Warfarin: A Trial Comparing Usual Care Warfarin Initiation to PerMIT Pharmacogenetic Guided Warfarin Therapy
Acronym: PerMIT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Robert Pendleton (Other)
Collaborators: University of Louisville (Other)
Responsible Party: Sponsor-Investigator, Robert Pendleton, Associate Professor of Clinical Medicine; Director Hospitalist Program; Medical Director Thrombosis Service, University of Utah
Organization: University of Utah (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 35279
Record Dates: First submitted 2009-10-08; First posted 2009-10-12 (Estimated); Results first posted 2013-05-16 (Estimated); Last update posted 2015-06-24 (Estimated); Status verified 2015-05

CONDITIONS: Blood Clotting
Keywords: Warfarin; Pharmacogenetic
MeSH Terms: conditions — Thrombosis | interventions — Warfarin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Warfarin, control (Active Comparator): Subjects naive to warfarin therapy with anticipated warfarin duration of at least 12 weeks managed by usual care dosing.
  Interventions: Drug: Warfarin
- Warfarin: PERMIT (Experimental): Subjects naive to warfarin therapy with anticipated warfarin duration of at least 12 weeks managed by warfarin pharmacogenetic dosing (warfarin dosing using genetic information incorporated into the PERMIT algorithm).
  Interventions: Genetic: warfarin pharmacogenetic dosing

INTERVENTIONS:
Genetic: warfarin pharmacogenetic dosing — Warfarin pharmacogenetic dosing incorporated into a validated clinical algorithm displayed in a computer (PERMIT) management interface
  Arms: Warfarin: PERMIT
Drug: Warfarin — Usual care warfarin dosing
  Arms: Warfarin, control

SUMMARY:
Warfarin is the most commonly used oral anticoagulant medicine (blood thinner). Although this medicine works well, it is difficult to know how much medicine a patient needs. Many things affect how much medicine a patient needs and doses can be very different from patient to patient. It is important for patients to get the right dose to prevent clotting or bleeding problems that can happen with this medicine if the dose is too low or too high. These problems can be life-threatening. To help find the right dose, patients on warfarin must have frequent blood tests to measure how well the medicine is working. The investigators know differences in people's genes can affect how much warfarin medicine someone needs, but they don't yet know with certainty how to use this information in making patient care decisions. The hypothesis of this study is that using a patients warfarin related genetic information incorporated into a computer algorithm to be used by a warfarin provider will lead to better warfarin management compared to usual care.

DETAILED DESCRIPTION:
Warfarin is the most commonly used oral anticoagulant medication. Due to the difficulty in determining an individual's proper warfarin dose, therapy is typically initiated with a standard dose followed by INR monitoring with frequent dose adjustment to ensure the medicine is working properly. Unfortunately, therapeutic warfarin doses vary significantly from patient to patient, so that even a standard dose can lead to excessive anticoagulation with its associated risk of causing life-threatening hemorrhaging. Genetic and non-genetic factors both influence an individual's warfarin dose requirement and response characteristics. There has been substantial evidence demonstrating a clear gene-dose relationship. Although this importance of pharmacogenetics to warfarin therapy is understood, clear guidance for how such information should be applied to patient therapy is woefully absent. The Personalized Medicine Interface Tool (PerMIT) is a software utility that supplies this critical guidance by modeling the dose requirements and response characteristics of individual patients based on their genotypic and physical characteristics. Using state-of-the-art multivariate computations, PerMIT calculates a warfarin maintenance dose estimate and also models the influence of repeated dosing on plasma drug concentration.

Both genetic and non-genetic factors (such as age, weight and gender) influence warfarin dose requirement and response characteristics of the individual. Recently, multi-variate mathematical equations, which take into account these genetic and non-genetic factors, such as age, weight and gender, have been developed to calculate an estimate of the warfarin maintenance dose requirement (Linder 2002, Zhu 2007, Sconce 2005, Millican 2007). The temporal response to routine administration of medications is dictated by the clearance rate of the medication and its effective concentration, the blood concentration over the dosing interval that is required to elicit the desired pharmacologic effect. The clearance of S-warfarin is primarily dictated by the patient's Cytochrome P4502C9 (CYP2C9) genotype, whereas the effective S-warfarin concentration is primarily dictated by the patient's vitamin K epoxide reductase complex protein 1 (VKORC1) genotype (Linder 2002, Herman 2005, Zhu 2007).

It is now well-known that genetic variants of CYP2C9 lead to decreased S-warfarin metabolism (clearance) and an increased elimination half-life. The elimination half-life of medications dictates the time required for repeated dosing to result in reproducible drug concentrations over the dosing interval for a given dosage. This situation is referred to as steady-state and is the most reliable time to interpret the dose-response relationship (INR measurements). S-warfarin half-life can be estimated based on the individual's CYP2C9 genotype (Linder 2002, Herman 2005, Loebstein 2001) and the steady-state concentration of S-warfarin under optimal anti-coagulation conditions is closely related to the patient's VKORC1 genotype (Zhu 2007).

PerMIT: Warfarin has clear theoretical benefits and has been demonstrated to be accurate; however, prospective randomized control clinical trials are required to demonstrate the efficacy of the PerMIT: Warfarin software in comparison to standard of care. We have designed this two-arm, prospective randomized control trial to directly assess the efficacy of PerMIT: Warfarin in (a) identifying patients' optimal dose requirements; (b) reducing patients' time to achieve stable therapy; (c) reducing the frequency of out-of-range INR measurements; and (d) reducing the number of dose adjustments. This study will evaluate whether, and to what degree, PerMIT: Warfarin improves these patient care outcomes and, by extension, reduces their risk of adverse drug reactions when compared to patients who receive therapy based on the standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Prescribed warfarin for any indication, so long as they are naïve to the drug at enrollment and are expected to receive therapy for at least 12 weeks

Exclusion Criteria:

* Recent cardiothoracic surgery as indication for warfarin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2009-08; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert C Pendleton, MD, Principal Investigator — University of Utah Health Care
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Twenty six subjects were enrolled and randomized
Pre-assignment Details: Naive to warfarin were randomized to groups
Groups:
- Warfarin: PERMIT: Subjects naive to warfarin therapy with anticipated warfarin duration of at least 12 weeks managed by genetic guided warfarin dosing incorporated into the PERMIT algorithm.
Period: Overall Study
Arm/Group | Warfarin, Control | Warfarin: PERMIT
Started | 13 | 13
Completed | 13 | 13
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Warfarin, Control | Warfarin: PERMIT | Total
Number analyzed (Participants) | 13 | 13 | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 5 | 11
  >=65 years | 7 | 8 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 45 (10) | 59 (10) | 52 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 12
  Male | 7 | 7 | 14
Region of Enrollment [Number; unit: participants]
  United States | 13 | 13 | 26

OUTCOME MEASURES:

1. Primary Outcome: The Number of Days to First International Normalized Ratio (INR) Within Therapeutic Range
Description: The number of days to first International Normalized Ratio (INR) is being measured from initiation of warfarin to the time when a subject first has an INR lab test result within +/- 0.5 of mean target INR range. The period during which this time interval could be measured is any time during the subject's warfarin therapy.
Time Frame: variable as defined
Population: analysis per protocol
Measure: Median (Standard Deviation); unit: days
Groups:
- Standard: Standard of care warfarin management
- PERMIT: Warfarin management with use of gene-based warfarin dosing algorithm
Arm/Group | Standard | PERMIT
Number analyzed (Participants) | 13 | 13
days | 8.3 (2) | 4.7 (2)

2. Secondary Outcome: Adverse Major and Minor Bleeding Events
Description: Number of major and minor bleeding events
Time Frame: 12 week
Measure: Number; unit: number of bleeding events
Arm/Group | Warfarin, Control | Warfarin: PERMIT
Number analyzed (Participants) | 13 | 13
number of bleeding events | 0 | 0

3. Secondary Outcome: Thrombotic Complication
Description: Number of thrombotic events
Time Frame: 12 week
Measure: Number; unit: number of thrombotic events
Arm/Group | Warfarin, Control | Warfarin: PERMIT
Number analyzed (Participants) | 13 | 13
number of thrombotic events | 0 | 0

ADVERSE EVENTS:
Arm/Group | Warfarin, Control | Warfarin: PERMIT
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/13
Other Adverse Events (participants affected / at risk) | 0/13 | 0/13

LIMITATIONS AND CAVEATS:
Small sample size in this pilot trial

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes